CLINICAL TRIAL: NCT02361632
Title: Does Adding Milk to Coffee Change Gastric Volume?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MK
Record Dates: First submitted 2015-01-28; First posted 2015-02-12 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Aspiration of Gastric Content
MeSH Terms: interventions — Coffee; Milk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Dietary Supplement. Participants drink coffee with or without milk in following order:
  1. Black coffee
  2. Coffee with 20% milk added
  3. Coffee with 50% milk added
  Interventions: Dietary Supplement: Coffee with or without milk
- Group 2 (Experimental): Dietary supplement. Participants drink coffee with or without milk in following order:
  1. Coffee with 20% milk added
  2. Black coffee
  3. Coffee with 50% milk added
  Interventions: Dietary Supplement: Coffee with or without milk
- Group 3 (Experimental): Dietary supplement. Participants drink coffee with or without milk in following order:
  1. Black coffee
  2. Coffee with 50% milk added
  3. Coffee with 20% milk added
  Interventions: Dietary Supplement: Coffee with or without milk

INTERVENTIONS:
Dietary Supplement: Coffee with or without milk — Intervention :30 participants were randomized to 3 Groups, 10 persons in each group. All participants fasted 6 hours for solid food before gastric volume was measured by Magnetic Resonance Imagining ( MRI). 2 hours before MRI examination, each participant ingested either 175 ml black coffee, 175 ml coffee with 20% milk or 175 ml coffee with 50% milk in the order defined for the group (arm).

SUMMARY:
The intention of this study is to determine wether coffee added milk change gastric volume in comparison with gastric volume after drinking black coffee

DETAILED DESCRIPTION:
Thirty participants - divided in tree groups - drink coffee with or without milk after six hours fast for solid food. Each group drinks both coffee with or without milk in different order. Two hours after drinking coffee gastric volume is measured by Magnetic Resonance Imagining.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Former or present gastric history, pregnancy, claustrophobia, metal implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in gastric volume after 175 ml coffee with 20% full fat milk compared with gastric volume after 175 ml black coffee . | "Up to 1 year" asses and proces

SECONDARY OUTCOMES:
Change in gastric volume after 175 ml coffee with 50% full fat milk compared with gastric volume after 175 ml black coffee | "Up to 1 year" asses and proces

CONTACTS AND LOCATIONS:
Overall Officials: Karin T Beier, MEd, Study Chair — Aarhus University Hospital Skejby

REFERENCES:
- [Derived] Larsen B, Larsen LP, Sivesgaard K, Juul S. Black or white coffee before anaesthesia?: A randomised crossover trial. Eur J Anaesthesiol. 2016 Jun;33(6):457-62. doi: 10.1097/EJA.0000000000000457. PMID 27035595